CLINICAL TRIAL: NCT04867681
Title: Study of the Impact on the Therapeutic Alliance of a Short Initial Psychoeducation Programme in Patients With Early Schizophrenia
Acronym: EPPICS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-AOI-06
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of a short psycho-education programme (Experimental)
  Interventions: Behavioral: Psycho-education programme
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Psycho-education programme — 4 individual sessions (S1, S2, S3, S4) of one hour each spread over 2 weeks, i.e. 2 sessions per week. S1 explains the different clinical signs and discusses the prognosis of the disease, S2 deals with the question of drug treatments, their different forms and their mechanisms of action. S3 discusses the evolution of the disease and the organisation of the care pathway. Finally, S4 looks at the aspects of quality of life, lifestyle and the fight against addictive co-morbidities, and concludes with a review of the patient's motivation and involvement in the subjects covered.
  Arms: Administration of a short psycho-education programme

SUMMARY:
Schizophrenia is a serious, disabling and unfortunately common disease. Its prevalence is in the order of 0.6 to 1% in the general population, a figure that remains relatively stable in the various cultures. The overall prognosis, particularly in terms of function, remains largely negative. The investigators know that a global management can considerably slow down this unfavourable evolution: according to the recommendations, the patient suffering from schizophrenia requires an effective and well-tolerated pharmacotherapy, associated with an adapted psychotherapy as well as cognitive remediation workshops, training in social skills, and psycho-education. There are indeed a large number of studies that have shown these elements in patients with schizophrenic disorders that have been present for several years. The investigators now know that early treatment is a key prognostic element. Indeed, the earlier care is provided during the first psychotic episode, the better the subsequent prognosis: the probability of further decompensation is reduced, as is the risk of developing deficits, such as cognitive difficulties. However, there is a lack of access to all the recommended aspects of management in the initial phase of the disorder, particularly concerning early psycho-educational programmes for patients, which have been relatively little studied in clinical research. In this context, it seems relevant to study the impact of a new programme of this type on a fundamental parameter, conditioning the subsequent access to care: the therapeutic alliance. "PPIC" is a short psycho-educational programme in 4 sessions, specifically designed to accompany young patients, and focused on the issues of this crucial period of the care process.

ELIGIBILITY:
Inclusion Criteria:

* French speaking
* Presenting a first or second acute psychotic episode, corresponding according to DSM 5 criteria to:

  * A brief psychotic disorder
  * And/or a schizophrenic disorder evolving for less than 2 years,
* Hospitalized in full time or in day care,
* Understanding and accepting the constraints of the study,

Exclusion Criteria:

* Patient under guardianship
* Patient participating in another study
* Patient in hospital under restraint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Therapeutic alliance scale | 3 months
  Mean change in the HAq-IIp therapeutic alliance score at 3 months after administration of the psycoeducation programme, compared between the active and control arms.
  This is a self-questionnaire evaluating the patient's subjective perception of his relationship with his therapist using 19 items, graded from 1 ("totally disagree") to 6 ("completely All right ").

CONTACTS AND LOCATIONS:
Overall Officials: Bruno GIORDANA, Dr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No